CLINICAL TRIAL: NCT02948413
Title: Exploring the Influence of Psychosocial Distress and Lifetime Trauma Exposure on Traumatic Stress Among Oncology Patients on Clinical Trials
Brief Title: Influence of Psychosocial Distress and Lifetime Trauma Exposure on Traumatic Stress Among Oncology Patients on Clinical Trials
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 170010; 17-CC-0010
Record Dates: First submitted 2016-10-27; First posted 2016-10-28 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Lymphoma; Mesothelioma; Prostate Cancer; Leukemia
Keywords: Traumatic Stress; Oncology; Lymphoma; Leukemia
MeSH Terms: conditions — Lymphoma; Mesothelioma; Prostatic Neoplasms; Leukemia; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group of patients with Cancer: Patients with cancer (lymphoma, leukemia, prostate cancer, and mesothelioma) on clinical trials at the NIH Clinical Center.

SUMMARY:
Background:

A cancer diagnosis is a threat to life and bodily integrity. This can cause people with cancer to experience traumatic stress. Researchers want to better understand the types of stress and emotional reactions people with cancer experience. They also want to know if the stress people with cancer have had during their life affects their stress related to cancer.

Objective:

To see if lifetime traumas, along with psychosocial distress, can predict traumatic stress symptoms in people with cancer.

Eligibility:

People ages 18 and older who have had or are currently getting care from the NIH Clinical Center for one of these cancers:

Leukemia

Lymphoma

Mesothelioma

Prostate cancer

Design:

Participants will be screened with name, date of birth, and diagnosis.

Participants will allow access to their medical records.

Participants will complete, online or in person, a demographic sheet and 3 questionnaires:

The PTSD Checklist for DSM-5: This assesses traumatic stress symptoms and takes 5 10

minutes to complete.

The Life Events Checklist for DSM-5: This assesses potentially traumatic life events and

takes about 5 minutes to complete.

The Brief Symptoms Inventory 18: This assesses psychosocial distress and takes about 4

minutes to complete....

DETAILED DESCRIPTION:
Background:

* The American College of Surgeons requires accredited cancer hospitals to screen for distress.
* Providers at the NIH CC do not uniformly screen for traumatic stress in oncology patients but have observed innumerable patients with deficits in social functioning, difficulty adhering to treatment, and trouble coping due to oncology related traumatic stress.
* A seminal distress study reported the prevalence of distress for 14 cancer diagnoses was as high as 43.4% with prevalence of distress in the 30% range for the diagnoses covered in this study.
* It has been shown that a cancer diagnosis represents a threat to life and bodily integrity and can create a sense of loss of social and occupational roles, causing one s adaptive capacity to become overwhelmed.
* In oncology patients, the literature reports that symptoms or traumatic stress range from 20% with early stage cancer to 80% in those with recurrent disease.
* The outcome of this study will provide information about traumatic stress, aid in the identification of it, and provide guidance on trauma informed care for this population.

Objectives:

* A descriptive study to explore the relationships between levels of psychosocial distress and levels of traumatic stress symptoms (TSS) in patients with cancer (lymphoma, leukemia, prostate cancer, and mesothelioma) on clinical trials at the NIH Clinical Center.
* We will also describe the relationship between psychosocial distress and TSS in the context of the number of lifetime traumas experienced by patients enrolled on a clinical trial at the NIH for cancer treatment.

Eligibility:

* Patients receiving treatment at the NIH CC will be recruited from four diagnostic groups: leukemia, lymphoma, mesothelioma, and prostate.
* Inclusion criteria include: diagnosed and treated for one of four types of cancer (patients can have any stage of one of these four types of cancer and can be at any point in the treatment continuum); aged 18 and over; able to understand and willing to sign a written informed consent document to participate in this study; enrolled in a clinical trial and actively followed on at the NIH CC.

Design:

* This study is an exploratory cross-sectional survey design.
* Data from the standardized measures (e.g. BSI-18, LEC-5, and the PCL-5) and demographic and medical history from the medical charts will describe the sample.
* Protocol participation is estimated to take approximately 10-15 minutes per patient.
* To address the primary objective, a backwards stepwise process will be used to identify covariate variables that will be used in the final model. This will allow for the data to present naturally occurring gaps in p-values to inform significance.
* Bi-variate analysis such as t-tests to compare means, time since diagnosis, time since clinical trials participation (e.g. treatment) and demographics, will be used to explore differences and relationships among the main variables and the demographic and illness-related variables.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study is open to all people with or who have been treated for cancer at the NIH CC in Bethesda, Maryland and meet the following criteria. This is done to provide the richest cross-section possible in this availability sample of patients undergoing or post treatment. Eligibility criteria include participants who are:

* Currently diagnosed or have been diagnosed with one of four types of cancer: leukemia, lymphoma, mesothelioma, and prostate cancer. Patients can have any stage of one of these four types of cancer and can be at any point in the treatment continuum, including active treatment, remission, recurrence, and surveillance or watchful waiting. An oncology diagnosis is considered sufficient for this protocol if it is sufficient for the patient to be enrolled in and actively followed on an oncology protocol at the NIH CC;
* Those who are pregnant are eligible to participate;
* Those who are HIV positive or have been diagnosed with AIDS in addition to carrying an oncology diagnosis are eligible to participate;
* Those who are aged 18 and over, as the research instruments have not been validated in individuals under the age of 18;
* Able to understand and willing to sign a written informed consent document to participate in this study;
* Enrolled in and actively followed on a clinical trial at the NIH CC.
* If applicable, agrees to complete study questionnaires on line.

EXCLUSION CRITERIA:

* Inability to meet the inclusion criteria;
* Inability to provide informed consent;
* Individuals with limited English proficiency as the research instruments have not been translated into or validated in languages other than English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is open to all people with or who have been treated for cancer at the NIH CC in Bethesda, Maryland and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Traumatic Stress Symptoms | Single Time Point
  A descriptive study to explore the relationships between levels of psychosocial distress and levels of traumatic stress symptoms (TSS) in patients with cancer (lymphoma, leukemia, prostate cancer, and mesothelioma) on clinical trials at the NIH Clinical Center.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Hendricks, Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gurevich M, Devins GM, Rodin GM. Stress response syndromes and cancer: conceptual and assessment issues. Psychosomatics. 2002 Jul-Aug;43(4):259-81. doi: 10.1176/appi.psy.43.4.259. PMID 12189252
- [Background] Cella DF, Mahon SM, Donovan MI. Cancer recurrence as a traumatic event. Behav Med. 1990 Spring;16(1):15-22. doi: 10.1080/08964289.1990.9934587. PMID 2322653
- [Background] Zabora J, BrintzenhofeSzoc K, Curbow B, Hooker C, Piantadosi S. The prevalence of psychological distress by cancer site. Psychooncology. 2001 Jan-Feb;10(1):19-28. doi: 10.1002/1099-1611(200101/02)10:13.0.co;2-6. PMID 11180574
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-CC-0010.html